CLINICAL TRIAL: NCT01642706
Title: Regulatory B Cells in Inflammatory Rheumatisms, Systemic Auto-immune Diseases in Adults and Biomarkers of Response to Biologic Treatments
Brief Title: Regulatory B Cells in Inflammatory Rheumatisms and Biomarkers of Response to Biologic Treatments
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: 8969
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis; Systemic Lupus Erythematosus; Sjogren's Syndrome; Scleroderma; Spondylitis; Gout; Spinal Disease; Chondrocalcinosis
Keywords: Regulatory B cells; Rheumatoid arthritis; Biomarker
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Lupus Erythematosus, Systemic; Sjogren's Syndrome; Scleroderma, Diffuse; Spondylitis; Gout; Spinal Diseases; Chondrocalcinosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Comparison of Bregs levels
  Lymphocytes will be analyzed from :
  * circulating blood
  * serum
  * articular serum
  * synovial membrane
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients: Patients affected by Rheumatoid arthritis.
- Control: Subjects affected by either :
  * mechanical pathology
  * systemic auto-immune pathology
  * other inflammatory rheumatism

SUMMARY:
B cells are known to play an important role in auto-immune diseases by activating T cells, secreting inflammatory cytokines and autoreactive antibodies. However, a sub-type of B cells named regulatory B cells or Bregs has recently shown capacities to prevent or cure arthritis in mouse models. Bregs have also been identified in humans.

DETAILED DESCRIPTION:
B cells are known to play an important role in auto-immune diseases by activating T cells, secreting inflammatory cytokines and autoreactive antibodies. However, a sub-type of B cells named regulatory B cells or Bregs has recently shown capacities to prevent or cure arthritis in mouse models. Bregs have also been identified in humans. Main objective: To study Bregs abnormalities in patients with rheumatoid arthritis (RA) at different stages of the disease compared to subjects with mechanical pathologies.Secondary objectives:- To evaluate the specificity of any abnormalities identified in RA by studying Bregs in patients with other autoimmune or other inflammatory joint diseases.- To evaluate the effect of biological and synthetic treatments on Bregs in patients with RA. - To assess whether the rate of Bregs before treatment is predictive of response to biological and synthetic treatments.

ELIGIBILITY:
Inclusion Criteria:

For RA patients and control patients:

* Age over 18 year old
* Blood sample taken as part of the usual management
* Steroid less than or equal to 15 mg/day and stable for at least a week

For RA patients:

* Patient with RA meeting the ACR / EULAR 2010

For control patients:

* Patients with systemic autoimmune disease (lupus, Sjogren's syndrome, scleroderma) or other inflammatory arthritis (spondylitis, crystals) or a mechanical pathology (limb osteoarthritis or spinal pathology) .

Exclusion Criteria:

* steroids over 15 mg/day
* rituximab infusion in less than 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and controls will be recruited in the Immuno-rheumatology Service of the University Hospital of Montpellier.
  They will be recruited during consultations or hospitalizations, when a blood sample is planned within the framework of their usual follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2012-07-02 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of Bregs levels | 30 months
  The levels of Bregs will be assessed in patients with RA and compared to subjects with mechanical pathologies.

SECONDARY OUTCOMES:
Change of Bregs levels after therapy | 30 months
  The levels of Bregs will be assessed in patients who will start a therapy within the framework of their usual follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Morel, MD, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Lapeyronie Hospital, Montpellier, France